CLINICAL TRIAL: NCT05240950
Title: A Clinical Study to Evaluate the Safety and Efficacy of Anti-CEA CAR-T Cells in the Treatment of Postoperative Minimal Residual Lesions in Colorectal Cancer Patients With Liver Metastases
Brief Title: Anti-CEA CAR-T Cells to Treat Colorectal Liver Metastases
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Wei Zhang, Director of Colorectal Surgery Department, Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHCRS-CEA CAR-T
Record Dates: First submitted 2021-12-26; First posted 2022-02-15 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Colorectal Cancer; Metastatic Liver Cancer
Keywords: colorectal cancer; liver metastasis; CAR-T cell; minimal residue disease
MeSH Terms: conditions — Colorectal Neoplasms; Liver Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRD or positive ctDNA patients to inject anti-CEA CAR-T cells (Experimental): Patients with liver metastasis of colorectal cancer after R0 surgery and adjuvant chemotherapy could not clear MRD (including patients with MRD still positive after the intermediate and final evaluation of adjuvant chemotherapy, and patients with MRD positive again after the end of adjuvant chemotherapy), and no measurable lesions or tumor remnants were found on imaging after surgery.
  Interventions: Drug: Anti-CEA CAR-T Cells

INTERVENTIONS:
Drug: Anti-CEA CAR-T Cells — The study will evaluate the safety of intravenous infusion of anti-CEA CAR-T (+) cells in humans at doses of 1×10^6/kg, 3×10^6/kg, and 6×10^6/kg using a standard "3+3" design and preliminarily observe the efficacy.

SUMMARY:
Recurrence of liver metastasis in colorectal cancer after R0 resection is mainly due to the invisible minimal residual disease, which are the main factors leading to metastasis and recurrence. Positive circulating tumor DNA (ctDNA) is the direct evidence of the minimal residual disease (MRD). In recent years, Chimeric Antigen Receptor T-Cell Immunotherapy (CAR-T) has made great breakthroughs, and has achieved good therapeutic effects in hematological tumors, but the research on solid tumors is limited. CEA expression is generally elevated in gastrointestinal tumors and is associated with high aggressiveness of tumors. At present, solid tumor cell therapy targeting CEA has been carried out at home and abroad, and has achieved certain efficacy. Anti-CEA CAR-T cells targeting CEA have been constructed in the pre-clinical study of this project, and the pre-clinical study results suggest good safety and effectiveness. Formation of minimal residual disease is associated with circulating blood in the residual tumor cells. Using this feature, this project intends to conduct a phase I clinical study on patients with minimal residual disease /positive ctDNA after R0 resection of colorectal cancer liver metastasis, so as to conduct preliminary exploration of anti-CEA CAR-T cell therapy, evaluate the safety and effectiveness of the therapy, determine the maximum tolerated dose (MTD), and provide guidance for subsequent drug dosage and clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old, ≤75 years old, male or female;
2. Patients diagnosed with liver metastasis of colorectal cancer underwent radical surgery for the primary lesion of colorectal cancer, and R0 resection was performed for the liver metastasis (R0 resection was required for other organ metastasis). There was no measurable disease or tumor remnants (except invisible or unmeasurable disease) were found by imaging examination after surgery;
3. Patients with CEA expression detected by immunohistochemistry in primary tumor and liver metastasis tumor tissues (CEA expression detected by pathology was more than 50%);
4. Life expectancy ≥6 months;
5. Performance status (PS) score 0-2, Karnofsky performance status (KPS) score above 60;
6. Patients with ctDNA MRD still positive or positive again after adjuvant chemotherapy (including preoperative neoadjuvant chemotherapy);
7. Important organ functions are sufficient, such as New York Heart Association (NYHA) heart function grade III or above, hemoglobin ≥90g/L, hypoxia; Liver function: total bilirubin ≤1.5×ULN (total bilirubin ≤3×ULN in liver metastasis), ALT≤2.5×ULN, AST≤2.5×ULN (ALT or/and AST≤5×ULN in liver metastasis); Renal function: serum creatinine ≤1.5×ULN and creatinine clearance rate ≥50 mL/min. The creatinine clearance rate was only calculated when serum creatinine ≤1.5×ULN. Minimum reserve of lung function (dyspnea no higher than grade 1 and oxygen saturation > 91% without oxygen);
8. Sufficient mononuclear cells (PBMC) can be obtained from peripheral veins without contraindications;
9. Patients of childbearing age had no birth plan within 1 year after cell infusion and took effective contraceptive measures.

Exclusion Criteria:

1. Have a history of severe central nervous system diseases;
2. Residual disease or tumor remnants can be seen in imaging, or tumor lesions cannot be resected in other tissues or organs;
3. The presence of serious non-malignant diseases, including autoimmune diseases, primary immunodeficiency diseases or obstructive or restrictive respiratory diseases;
4. Prior treatment with CAR-T or other gene-modified T cells;
5. Participated in other clinical studies within 30 days prior to screening or plan to participate in other clinical studies during the study period;
6. Patients with active Hepatitis B (HBV-DNA copy number >105copies/ml), active Hepatitis C (HCV-RNA copy number >ULN), HIV infection, treponema pallidum infection at screening time;
7. The existence of uncontrollable systemic infectious diseases;
8. Other multiple malignant tumors in addition to colorectal cancer and its metastasis;
9. Chinese herbal medicine, systemic glucocorticoids or other immunosuppressants may be required within 2 weeks prior to enrollment or during the trial period, which may negatively affect lymphocyte activity or number;
10. Pregnancy and lactation;
11. The existence of severe gastroduodenal ulcer, severe ulcerative colitis and other serious intestinal inflammation;
12. The existence of serious respiratory diseases;
13. Those who cannot provide enough white tablets for tumor pathology for next-generation sequencing (NGS) detection (at least 3 white tablets are expected);
14. The investigator judged that there were other conditions that were not suitable for the clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-08-25 (Estimated); Primary Completion 2023-12-25 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
Security (Incidence and severity of adverse events) | Observation 28 days after CAR-T cells infusion
  To evaluate the possible reatment related adverse events(TEAEs) occurred within the first 28 days after anti-CEA CAR-T infusion, including replicative lentiviruses(RCL), anti-drug antibody(ADA), and the incidence and severity of symptoms such as cytokine release syndrome(CRS) and CAR-T related encephalopathy syndrome(CRES).
Effectiveness (minimal residual disease) | 24 months after R0 resection
  Recurrence by ctDNA MRD detection or imaging diagnosis
Efficacy (recurrence-free survival) | 2 years after CAR-T cells infusion
  2-year recurrence-free survival rate based on imageological examination.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) indicator (Cmax) | 2 years after CAR-T cells infusion
  The peak concentration of anti-CEA CAR-T cells amplified in the peripheral blood (Cmax, detected by flow cytometry and qPCR).
Pharmacokinetics (PK) indicator (AUC) | 2 years after CAR-T cells infusion
  The exposed quantity of anti-CEA CAR-T cells amplified in the peripheral blood(aera under the curve, AUC, detected by flow cytometry and qPCR).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Colorectal Surgery in Changhai Hospital, Shanghai, Shanghai Municipality, China